CLINICAL TRIAL: NCT04434859
Title: Incidence of Temporomandibular Disorders Among Patients With Tinnitus
Brief Title: Temporomandibular Disorders Among Patients With Tinnitus
Acronym: TMDTIN
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 256-20
Record Dates: First submitted 2020-06-10; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Tinnitus; Temporomandibular Disorder
MeSH Terms: conditions — Tinnitus; Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with tinnitus: Patients (over 18 years old) seen at the medical center due to tinnitus, lasting at least 3 months.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The incidence of temporomandibular disorders will be studied among patients with tinnitus, by the use of patient's history and physical examination.

DETAILED DESCRIPTION:
The patients with tinnituswill be asked about symptoms related to temporomandibular disorders, and also will be examined in order to diagnose such disorders.

ELIGIBILITY:
Inclusion Criteria:

* Tinnitus lasting more than 3 months

Exclusion Criteria:

* Head and Neck Space Occupying Lesion
* Previous degenerative disease of the temporomandibular koint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with tinnitus lasting more than 3 months
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Description of temporomandibular disorders in the patient's history | 1 year
  A questioannaire asking specifically about pain in the tempromandibular joint, headaches, clicks, tempromandibular joint locking and dislocation
Positive findings in the physical examination of the temporomandibular joint and muscles | 1 year
  The following parameters will be documented: clicks, maximal opening of the mouth, signs of teeth grinding, tenderness on the mastication muscles

IPD SHARING:
Plan to Share IPD: No